CLINICAL TRIAL: NCT01543490
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Parallel-Group, Comparative Study to Evaluate the Clinical Efficacy and Safety of ISV-305 (0.1% Dexamethasone) Compared to Vehicle in the Treatment of Subjects With Blepharitis
Brief Title: Comparative Study to Evaluate ISV-305 Compared to Vehicle in Blepharitis Subjects
Acronym: ISV-305
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-12-305-001
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Active, Symptomatic Blepharitis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ISV-305 (Experimental): 0.1% dexamethasone in DuraSite® 2
  Interventions: Drug: ISV-305
- Vehicle (Placebo Comparator): DuraSite® 2 vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: ISV-305 — Dexamethasone in DuraSite® 2 twice daily for 2 weeks
  Arms: ISV-305
Other: Vehicle — Vehicle twice daily for 2 weeks
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of ISV-305 (Dexamethasone in DuraSite® 2) compared to Vehicle in the treatment of subjects with active, symptomatic Blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 1 years of age and have a clinical diagnosis of active, symptomatic blepharitis
* Signature of the subject or parent(s) or legally authorized representative on the Informed Consent Form, and when appropriate the minor's assent in accordance with local regulations
* Are willing and able to follow all instructions and attend all study visits (this applies to parent or caregiver for subjects too young to self-apply investigational product)
* Are willing to avoid disallowed medication for the duration of the study
* If female is of childbearing potential, agree to and submit a urine sample for pregnancy testing (prior to enrollment and at the end of the study) and use effective contraception for the duration of the study
* Male subjects whose female partners are not post-menopausal must agree to one of the following: 1) completely abstain from sexual intercourse, 2) use a barrier method (condoms) with spermicide during sexual intercourse for the duration of the study, 3) provide documentation for having had a vasectomy (with documented infertility)
* Additional inclusion criteria also apply

Exclusion Criteria:

* Have known sensitivity or poor tolerance to any component of the study drugs
* Have had eyelid surgery in the study eye within twelve (12) months prior to Visit 1 or plan to have eyelid surgery during the study
* Have an acute ocular infection (bacterial, viral or fungal) or active ocular inflammation other than blepharitis in the study eye
* Have used topical medications on the eyelids or topical ophthalmic corticosteroid medications or systemic use of a corticosteroid mediation within 14 days prior to dosing and/or plan to use them throughout the duration of the study
* Be currently pregnant, nursing, or planning a pregnancy; or be a woman who has a positive urine pregnancy test
* Have prior (within 30 days prior to dosing) or anticipated concurrent use of an investigational drug or device
* Have a condition or a situation which, in the investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation
* Additional exclusion criteria also apply

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ISV-305: ISV-305 was administered as a topical ophthalmic formulation of 0.1% dexamethasone in DuraSite® 2 vehicle (InSite Vision's drug delivery system) twice daily (one drop in the morning and one drop in the evening) for 14 days.
- Vehicle: Vehicle (DuraSite® 2 vehicle) was administered as a matching topical ophthalmic formulation without dexamethasone twice daily (one drop in the morning and one drop in the evening) for 14 days.
Period: Overall Study
Arm/Group | ISV-305 | Vehicle
Started | 368 | 190
Completed | 352 | 185
Not Completed | 16 | 5
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lack of Efficacy | 3 | 3
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other-Various Administrative Reasons | 1 | 2

BASELINE CHARACTERISTICS:
Population: Demographics were summarized for the Intent-to-treat (ITT) Population, which included all randomized participants regardless of whether post-baseline measures were collected or study treatment was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-305 | Vehicle | Total
Number analyzed (Participants) | 368 | 190 | 558
Age, Customized [Count of Participants; unit: Participants]
  < 17 years | 0 | 0 | 0
  17 to < 65 years | 146 | 66 | 212
  ≥ 65 years | 222 | 124 | 346
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 107 | 316
  Male | 159 | 83 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or Black | 20 | 2 | 22
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  White | 334 | 184 | 518
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Mixed | 1 | 0 | 1
  Other | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 368 | 190 | 558

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the ITT Population With a Reduction in the Day 1 (Baseline) Total Clinical Signs and Symptom Score by at Least 2 Units at Day 15 With No Worsening of Any Sign or Symptom
Description: The clinical signs of blepharitis (eyelid swelling, eyelid redness, eyelid debris) were evaluated at every visit and scored by the investigator using a 0 to 3 grading scale (in general 0 = none, 1 = mild, 2 = moderate, and 3 = severe). The symptom of eyelid irritation was also evaluated at every visit and graded by the participant using a 0 to 3 grading scale (0 = almost none of the time - ≤ 25% of the time, 1 = occasionally - 26-50% of the time, 2 = frequently - 51-75% of the time, 3 = almost all of the time - ≥ 76% of the time). For each visit, the total clinical signs and symptom score was obtained by adding each of the individual scores for each domain (eyelid swelling, eyelid redness, eyelid debris, and eyelid irritation). Participants with a decrease in total clinical signs and symptom score at Day 15 by at least 2 units from Day 1 (baseline) with no increase in any sign and symptom were defined as Responders, and those not meeting these criteria were defined as Non-responders.
Time Frame: Day 15
Population: ITT Population, which included all randomized participants regardless of whether post-baseline measures were collected or study treatment was received. The participants only with valid measurement at Day 15 were used as the denominator for percentages (353 out of 368 participants for ISV-305 and 185 out of 190 participants in Vehicle).
Measure: Count of Participants; unit: Participants
Arm/Group | ISV-305 | Vehicle
Number analyzed (Participants) | 353 | 185
Participants
  Responders | 276 | 129
  Non-responders | 77 | 56
Statistical Analysis 1: Comparison: ISV-305 vs Vehicle; Test type: Superiority — Statistical hypotheses testing for the primary efficacy endpoint was 2-sided and performed using a significance (alpha) level of 0.05; p = 0.0354, Fisher Exact — The p-value was from a 2-sided Fisher's exact test; The point estimate of treatment effect (ISV-305 compared with Vehicle) was reported using Fisher's exact test; Risk Difference (RD) = 8.5, 95% CI 2-sided [0.2 to 16.6], Standard Error of Mean 4.03 — The risk difference was obtained by taking the difference in proportions (ISV-305 minus Vehicle). A 2-sided exact unconditional 95% confidence interval (CI) was calculated

2. Secondary Outcome: Number of Participants With Complete Resolution of Eyelid Irritation (Last Observation Carried Forward [LOCF]) on Day 15 in ITT Population
Description: Complete resolution of eyelid irritation, which was defined as eyelid irritation with grading of 0, at Day 15 was analyzed. The symptoms of eyelid irritation were graded by the participant using a 0 to 3 grading scale, where 0 = almost none of the time - ≤ 25% of the time, 1 = occasionally - 26-50% of the time, 2 = frequently - 51-75% of the time, 3 = almost all of the time - ≥ 76% of the time.
Time Frame: Day 15
Population: ITT Population, which included all randomized participants regardless of whether post-baseline measures were collected or study treatment was received. Participants with a valid post-baseline measurement on or before at Day 15 were used as the denominator for percentages (368 for ISV-305 and 190 for Vehicle).
Measure: Count of Participants; unit: Participants
Arm/Group | ISV-305 | Vehicle
Number analyzed (Participants) | 368 | 190
Participants
  With Complete Resolution | 127 | 52
  Without Complete Resolution | 241 | 138
Statistical Analysis 1: Comparison: ISV-305 vs Vehicle; Test type: Superiority — Statistical hypotheses testing for the secondary efficacy endpoint was 2-sided and performed using a significance (alpha) level of 0.05, and missing data imputed using the LOCF approach; p = 0.1036, Fisher Exact — The p-value was from a 2-sided Fisher's exact test; The point estimate of treatment effect (ISV-305 compared with Vehicle) was reported using Fisher's exact test; Risk Difference (RD) = 7.1, 95% CI 2-sided [-1.3 to 15.0], Standard Error of Mean 4.07 — The risk difference was obtained by taking the difference in proportions (ISV-305 minus Vehicle). A 2-sided exact unconditional 95% CI was calculated

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the date of signing the consent form to the date of completion of the participant's final visit (Day 29). Ongoing AEs were followed beyond the final study visit at the discretion of the investigator, observed up to 41 days.
Description: Treatment-emergent adverse events were summarized for the Safety Population, which included all randomized participants who received at least one dose of study treatment (i.e., 367 and 188 participants in the ISV-305 and Vehicle arms, respectively).
Arm/Group | ISV-305 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/367 | 0/188
Serious Adverse Events (participants affected / at risk) | 4/367 | 0/188
Other Adverse Events (participants affected / at risk) | 7/367 | 5/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-305 (N=367) | Vehicle (N=188)
Syncope (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-305 (N=367) | Vehicle (N=188)
Conjunctival hyperaemia (Eye disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT01543490/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT01543490/SAP_000.pdf